CLINICAL TRIAL: NCT00264056
Title: Evaluation of the Safety and Efficacy of Systemic Chemotherapy Combined With Regional Hypothermia in Advanced Malignant Melanoma Patients With Locally Inoperable Progressive Soft Tissue Metastases
Brief Title: Efficacy of Chemotherapy Combined With Regional Hypothermia in Advanced Malignant Melanoma Patients With Progressive Soft Tissue Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fachklinik Hornheide an der Universität Münster (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOT-100
Record Dates: First submitted 2005-12-08; First posted 2005-12-12 (Estimated); Last update posted 2005-12-12 (Estimated); Status verified 2005-11

CONDITIONS: Advanced Metastastic Malignant Melanoma; Refractory to First-Line Chemotherapy Irresectable Progressive Soft Tissue Metastases
Keywords: malignant melanoma; hyperthermia; chemotherapy
MeSH Terms: conditions — Melanoma; Hyperthermia | interventions — Diathermy

INTERVENTIONS:
Device: hyperthermia

SUMMARY:
The incidence of malignant melanoma continues to rise throughout the world. Approximately 12 in 100,000 Germans are diagnosed with malignant melanoma per year. Malignant melanoma is often very aggressive since it may spread both through the lymphatic system and the bloodstream at an early stage of disease.

While treatment of localized disease is mostly surgical, in patients with extensive disease, prognosis remains poor; the primary standard therapy of metastastic disease comprises dacarbazine (DTIC) eventually combined with other chemotherapeutic agents e.g., cisplatin or BCNU. The duration of response to systemic chemotherapy is generally short and so far, no standard second-line treatment has been established.

To study the potential additional therapeutic effects of regional hyperthermia in advanced malignant melanoma patients with progressive chemotherapy refractory soft tissue metastases, in the present trial, we sought to compine local hyperthermia with concomitant systemic second-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70
* histologically proven malignant melanoma with advanced inoperable soft tissue metastases
* progressive disease upon systemic first-line chemotherapy
* 2 or more bidimensionally measurable soft tisue lesions
* WHO performance status (ECOG) of 2 or more
* life expectancy of 8 weeks and more
* prior informed consent

Exclusion Criteria:

* participation in other therapy studies
* pregnancy or breast feeding
* concomitant clinically significant infection
* cardiac pacemaker or other medical implants, or implants within the hyperthermia treated region (including a safe distance of 5 cm)
* lack of physiological heat sensitivity within the hyperthermia treated region (including a safe distance of 5 cm)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26
Dates: Start 2005-12; Study Completion 2007-06

CONTACTS AND LOCATIONS:
Overall Officials: Jens Atzpodien, MD, PhD, Principal Investigator — Fachklinik Hornheide an der Universität Münster
Locations (1):
- Fachklinik Hornheide at the University of Münster, Germany, Münster, Germany